CLINICAL TRIAL: NCT04219657
Title: Comparison of Outcome of Mesenchymal Stem Cells And Skin Graft With Skin Graft In Management of Traumatic Heel Pad Injuries of Children
Brief Title: Comparison Between Skin Graft Versus Skin Graft and Stem Cell Application
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sushil_Rijal
Record Dates: First submitted 2019-12-28; First posted 2020-01-07 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Accidental Wound; Heel Injury; Stem Cell Transplant
Keywords: spoke wheel injury; umbilical cord mesenchymal stem cells; skin grafting

STUDY DESIGN:
Intervention Model Description: Cases were divided into two groups. Group A included cases with skin graft only and group B included cases with skin graft and application of mesenchymal stem cells. Every odd patients were kept in group A and every Even patients were kept in group B.
Who Masked: Participant
Masking Description: cases included in study were randomly divided into two group. patients were masked about group. Every odd patients were kept in group A and every Even patients were kept in group B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skin grafting only (Experimental): All the cases in this group are managed with skin grafting only. Every odd case are kept in skin grafting only group.
  Interventions: Biological: mesenchymal stem cell application
- skin grafting and stem cell group (Experimental): All the cases in this group are managed with skin grafting and application of stem cells. every even cases are kept in skin grafting and stem cells group.
  Interventions: Biological: mesenchymal stem cell application

INTERVENTIONS:
Biological: mesenchymal stem cell application

SUMMARY:
Trauma is the leading cause of soft tissue loss of the heel. Children constitute the largest group of victims of such injuries. Spoke wheel injury, road traffic accident are common mode in the children. Oestern and Tscherne have classified soft tissue injuries into four grades from 0-4. The treatment of Grade 0 and 1 injuries is typical cleansing and application of a moist wound healing dressing. But further grades need surgical management with debridement and reconstruction. Grade III and IV can be reconstructed by using graft, flaps or various other techniques. . Skin grafting offers poor functional and cosmetic results, although it is commonly performed with good take rates. mesenchymal stem cells will be isolated from umbilical cord with informed consent from the mothers. This study will open a new avenue for the treatment of heel pad injury. . Since the use of stem cell (especially in Pakistan) is completely a new technique in the management of heel pad injury, it will provide insight for better management by accelerating the wound healing process.

DETAILED DESCRIPTION:
Trauma is the leading cause of soft tissue loss of the heel. Children constitute the largest group of victims of such injuries. Spoke wheel injury, road traffic accident are common mode in the children. These injuries can range from simple minor abrasions, lacerations to crushing of heel. Injury to heel pad and flap has serious impact in day to day life, causing disability because it is the major weight bearing area and inherently lacks adequate soft tissue.

Management of injury of heel pad in children depends on severity and extent of soft tissue injury. Oestern and Tscherne have classified soft tissue injuries into four grades from 0-4. The treatment of Grade 0 and 1 injuries is typical cleansing and application of a moist wound healing dressing. But further grades need surgical management with debridement and reconstruction.

Grade III and IV can be reconstructed by using graft, flaps or various other techniques. Simple skin graft, lateral rotational skin flap, local muscle flaps, ingenious fasciocutaneous island flaps, cross-leg or cross foot flap, free tissue transfer and staged or distant jumped flaps are historically included in reconstructive ladder in repairing these soft tissue injuries. Generally, free flap reconstruction is the ultimate step of degloving wound coverage. Despite availability of various reconstructive techniques, covering of soft tissue loss of heel in traumatic events, remains a difficult and demanding procedure, especially when it is associated with fractures and complex wounds. Skin grafting offers poor functional and cosmetic results, although it is commonly performed with good take rates.

Stem cells are potential alternative to promote cutaneous wound healing because of its unique features like self-renewal and differentiation capacity. Mesenchymal stem cells are type of adult stem cells that reside in various tissues of the body. Besides, these cells are preferred for cell based therapies because they have immunomodulatory properties. These cells can be isolated from bone marrow, adipose tissue and human umbilical cord blood and tissue. Recently,umbilical cord derived mesenchymal stem cells have shown a tremendous potential for use in tissue engineering and regenerative medicine. Previous studies indicate that these mesenchymal stem cells can accelerate wound healing by enhanced proliferation and migration of human fibroblast, enhancing secretion of elastin, synthesizing collagen, angiogenesis and further maturing blood vessels present in wound site. Stem cell-based therapies will definitely be the major part of clinical medicine in next decade.

In the current study, mesenchymal stem cells will be isolated from umbilical cord with informed consent from the mothers. This study will open a new avenue for the treatment of heel pad injury. Considering the role of stem cells in wound healing, study has been designed to accelerate the wound healing process in children with heel pad injury. Since the use of stem cell (especially in Pakistan) is completely a new technique in the management of heel pad injury, it will provide insight for better management by accelerating the wound healing process, reducing the hospital stay and cost of treatment. Rationale of our study aims to compare outcome of heel pad injury managed with skin graft with infiltration of mesenchymal stem cell Versus management with skin graft only.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric age group population (less than 12 years) irrespective of sex.
* Children with traumatic heel pad injury requiring skin grafting admitted through outdoor and emergency department.

Exclusion Criteria:

* Children with traumatic heel pad injury associate with other systemic injury requiring surgical/medical treatment other than skin graft/flap.
* Traumatic heel pad injury with calcaneal fracture.
* Children with traumatic heel pad injury with osteomyelitis, Idiopathic thrombocytopenic purpura, diabetes mellitus and immunodeficiency state under medication.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2016-10-29 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
Ranges of Movement of ankle joint | at 1st week of intervention and after at 12 weeks
  Average Ranges of Motion of ankle joint as described by American Academy of Orthopedic Surgeons is Dorsiflexion 0-20 degrees and Plantarflexion 0-50 degrees. In our scoring system dorsiflexion upto20 degree will be given 5 score and 0 degree will be given 0 score. Similarly, plantar flexion beyond 40 degree will be given 5 and 0 degree will be given 0 score.

SECONDARY OUTCOMES:
duration of hospital stay | from the date of admission to 2 weeks post admission
  Hospital stay will be measured in terms of duration from date of admission to date of discharge from ward. The average hospital stay of children with heel pad injury with skin grafting is one month in pediatric surgery department in Mayo hospital, King Edward Medical University. In our study wound healing will be said better if hospital stay after skin graft/ flap with stem cell application will be less than one month.
Weight bearing capacity of patients | at 1st week of intervention and after at 12 weeks
  Early weight bearing will be evaluated by pain intensity. Pain Score in this study will be measured by using Visual analogue scale (VAS). (Annex- 2) This scale is a valid tool for the measurement of pain intensity which has been widely used in diverse pediatric population. The scale is a continuous scale comprised of a horizontal or vertical line, usually 10 cm (100mm) in length, which is anchored by two extremes-no pain and worst possible pain. This scale is completed by treating consultant surgeon. Based on the distribution of visual analogue scale score in post-surgical patients, pain intensity is further classified as no pain, mild pain, moderate pain or severe pain with the cut points of 04mm, 5-44mm, 45-74mm and 75-100mm respectively.

CONTACTS AND LOCATIONS:
Overall Officials: FATIMA NAUMERI, assoc Prof, Study Director — King Edward Medical University
Locations (1):
- Pediatric Surgery Department, King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalam M, Faruquee S, Rahman S, Uddin H. Reconstruction of Heel: Options and Strategies. Bangladesh Journal of Plastic Surgery. 2010;1(1):14-8.
- [Background] Gupta H, Shrestha R. Bicycle-spoke injuries of the foot and ankle: A prospective study. Journal of College of Medical Sciences-Nepal. 2014;9(4):36-9.
- [Background] Aslam MR, Khan AS, Pasha IF, Taj RU. Reconstruction of hind foot defects. Professional Medical Journal. 2013;20(4):606-16.
- [Background] Lasanianos NG, Kanakaris NK. Soft Tissue Injuries. Trauma and Orthopaedic Classifications: Springer; 2015. p. 481-5
- [Background] Meland NB. Microsurgical reconstruction: the weightbearing surface of the foot. Microsurgery. 1990;11(1):54-8. doi: 10.1002/micr.1920110111. PMID 1970110
- [Background] Lim H, Han DH, Lee IJ, Park MC. A Simple Strategy in Avulsion Flap Injury: Prediction of Flap Viability Using Wood's Lamp Illumination and Resurfacing with a Full-thickness Skin Graft. Arch Plast Surg. 2014 Mar;41(2):126-32. doi: 10.5999/aps.2014.41.2.126. Epub 2014 Mar 12. PMID 24665420
- [Background] Fathi HR, Fathi M, Javid MJ. S-shaped reverse sural flap for reconstruction of tissue defect on heel. Burns Trauma. 2013 Jun 18;1(1):39-43. doi: 10.4103/2321-3868.113334. eCollection 2013. PMID 27574621
- [Background] Rodriguez J, Boucher F, Lequeux C, Josset-Lamaugarny A, Rouyer O, Ardisson O, Rutschi H, Sigaudo-Roussel D, Damour O, Mojallal A. Intradermal injection of human adipose-derived stem cells accelerates skin wound healing in nude mice. Stem Cell Res Ther. 2015 Dec 8;6:241. doi: 10.1186/s13287-015-0238-3. PMID 26645735
- [Background] Isakson M, de Blacam C, Whelan D, McArdle A, Clover AJ. Mesenchymal Stem Cells and Cutaneous Wound Healing: Current Evidence and Future Potential. Stem Cells Int. 2015;2015:831095. doi: 10.1155/2015/831095. Epub 2015 May 27. PMID 26106431
- [Background] Zhang J, Guan J, Niu X, Hu G, Guo S, Li Q, Xie Z, Zhang C, Wang Y. Exosomes released from human induced pluripotent stem cells-derived MSCs facilitate cutaneous wound healing by promoting collagen synthesis and angiogenesis. J Transl Med. 2015 Feb 1;13:49. doi: 10.1186/s12967-015-0417-0. PMID 25638205